CLINICAL TRIAL: NCT00910533
Title: Clinical and Microbiological Parameters in Patients With Early Lyme Neuroborreliosis
Brief Title: Study on Early Lyme Neuroborreliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Franc Strle, M.D., PhD, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LNB-0509
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2017-05

CONDITIONS: Nervous System Lyme Borreliosis
Keywords: Lyme neuroborreliosis
MeSH Terms: conditions — Lyme Neuroborreliosis | interventions — Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Lyme neuroborreliosis patients (Active Comparator)
  Interventions: Drug: ceftriaxone
- control subjects (No Intervention): Control subjects without a history of Lyme borreliosis.

INTERVENTIONS:
Drug: ceftriaxone — ceftriaxone 2 g od i.v. for 14 days
  Arms: Early Lyme neuroborreliosis patients

SUMMARY:
The purpose of this study is to determine clinical course and the sequelae of early Lyme neuroborreliosis after treatment with ceftriaxone.

ELIGIBILITY:
Inclusion Criteria:

* erythema migrans within 4 months before neurologic involvement and pleocytosis in patients >15 years old

Exclusion Criteria:

* pregnancy
* lactation
* history of adverse reaction to a beta-lactam antibiotic

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01-01; Primary Completion 2018-12-31 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Objective sequelae and post-treatment subjective symptoms in patients treated with ceftriaxone for early Lyme neuroborreliosis | 1 year follow-up

SECONDARY OUTCOMES:
Comparison of subjective symptoms between patients treated with ceftriaxone for early Lyme neuroborreliosis and control subjects without a history of Lyme borreliosis | 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD, Study Chair — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia